CLINICAL TRIAL: NCT03791567
Title: Expanded Access to Donislecel for Treatment Use
Brief Title: Islet Transplantation in Type I Diabetic Patients Using the University of Illinois at Chicago (UIC) Protocol
Status: Approved for marketing | Type: Expanded Access
Sponsor: CellTrans Inc. (Industry)
Responsible Party: Principal Investigator, Jose Oberholzer, Adjunct Professor of Surgery, University of Illinois at Chicago
Other Study IDs: EA IND11807-2007-0330
Record Dates: First submitted 2018-12-31; First posted 2019-01-02 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1; Type 1 Diabetes Mellitus; Islets of Langerhans Transplantation; Allogeneic Islet transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Transplantation

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Donislecel (allogeneic islets of Langerhans for transplant) — Intervention Description: The drug product consists of allogeneic human islets of Langerhans (islets) in serum-free transplant medium (indicator-free CMRL 1066 medium with HEPES, without sodium bicarbonate and supplemented with human albumin).

SUMMARY:
A Phase 3 clinical trial has been completed and demonstrated the safety and efficacy of allogeneic islet transplantation in improving glycemic control in Type 1 diabetic patients using the UIC protocol.The objective in offering expanded access to donislecel (allogeneic islets of Langerhans for transplant; IND BB-11807) for the treatment of brittle T1D is to bridge the gap between completed clinical trials and marketing (i.e. approval by the FDA of a biological license application). Expanded access will allow clinical trial subjects, as well as patients outside a clinical trial, to receive treatment. New patients participating in the expanded access protocol are required to meet exclusion and inclusion criteria.

DETAILED DESCRIPTION:
Expanded access to donislecel (allogeneic islets of Langerhans for transplant; IND BB-11807) is for the treatment of brittle T1D. Brittle T1D is a distinct subset of T1D, representing the most severe and difficult to manage manifestation of the disease. Standard therapies (i.e. exogenous insulin injections and insulin pumps) are not sufficient to regulate blood glucose levels for this subset of patients. Thus, the severity of disease and the lack of metabolic control that occur despite intensive insulin therapy in brittle T1D patients defines a patient population whose risk-benefit profile makes them suitable for islet transplantation. Eligible patients may receive one or several allogeneic pancreatic islet transplants. An independent Data Monitoring Committee (DMC), composed of 3 members who have training in medicine and/or organ transplantation, will review eligibility and safety data within 2 weeks after each islet transplantation and every two months thereafter. An independent monitor, who is knowledgeable about Good Clinical Practice (GCP) guidelines and regulations, monitors the study for compliance with 21 CFR and according to ICH GCP Guidelines. The UIC Institutional Review Board (IRB) reviews safety data annually and on occurrence of serious adverse events. The principal investigator also reports serious adverse events to the US Food and Drug Administration (FDA). Success, partial success, and failure criteria will be the same as indicated in the Phase III clinical trial. Patients will be closely monitored post-transplant by the UIC clinical team and/or their primary care physician for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must have Type 1 diabetes mellitus for more than 5 years, complicated by the following situations that persist despite intensive insulin management efforts:
* At least one episode of severe hypoglycemia in the past 3 years defined as an event with symptoms compatible with hypoglycemia in which the subject required the assistance of another person, and which was associated with either a blood glucose level < 50 mg/dL (2.8 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration
* Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at capillary glucose levels of < 54 mg/dL (3 mmol/L) as reported by the subject

Exclusion Criteria:

* Diagnosis of co-existing cardiac disease characterized by any one of these conditions:

  * Recent myocardial infarction (within past six months), or
  * Angiographic evidence of non-correctable coronary artery disease, or
  * Evidence of ischemia on functional cardiac exam (with a stress echo test recommended
  * for subjects with a history of ischemic disease).
  * Heart failure > New York Heart Assoication (NYHA) II
* Active alcohol or substance abuse-includes cigarette smoking (must be abstinent for six months). Active alcohol abuse should be considered using the current National Institute on Alcohol Abuse and Alcoholism (NIAAA) definitions.
* Psychiatric disorder making the subject not a suitable candidate for transplantation, e.g., schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medication. (A psychological or psychiatric consultation is required only if considered necessary by some current indication or history.)
* History of non-adherence to prescribed regimens
* Active infection including hepatitis C, hepatitis B, HIV
* TB (by history or currently infected as evidenced by a positive QuantiFERON® -TB Gold test or under treatment for suspected TB)
* Any history of malignancies except squamous or basal skin cancer. Any subject found to have squamous or basal cancer is required to have it removed prior to transplant.
* History of stroke within the past 6 months
* Body Mass Index (BMI) > 27 kg/m2.
* C-peptide response to glucagon stimulation (1 mg i.v.) (any C-peptide ≥ 0.3 ng/mL)
* Inability to provide informed consent
* Age less than 18 or greater than 65 years
* Creatinine clearance < 80 mL/min/1.73 m2 by 24-hour urine collection. If corrected creatinine clearance is < 80 and serum creatinine is < 1.2 mg/dl, then a nuclear renal scan is required to determine gomerular filtration rate.
* Serum creatinine consistently > 1.5 mg/dL
* Macroalbuminuria (urinary albumin excretion rate > 300 mg/24h)
* Baseline Hb < 12 gm/dL in women or < 13 gm/dL in men
* Baseline liver function tests (LFT) outside of normal range (An initial LFT test panel with any values > 1.5 times normal upper limits will exclude a subject without a re-test. A re-test for any values between normal and 1.5 times normal should be made, and if the values remain elevated above normal limits, the subject will be excluded.)
* Untreated proliferative retinopathy
* Positive pregnancy test, intent for future pregnancy, or male subjects' intent to procreate, unwilling to follow effective contraceptive measures, or presently breast-feeding
* Insulin requirement > 0.7 IU/kg/day
* HbA1c > 12%
* Hyperlipidemia (fasting LDL cholesterol > 130 mg/dL, treated or untreated; and/or fasting triglycerides > 200 mg/dL)
* Under treatment for a medical condition requiring chronic use of steroids other than a previous organ transplant
* Use of coumadin or other antiplatelet or anticoagulant therapy, or subject with PT INR > 1.5. Low dose aspirin is allowed after transplantation.
* History of Factor V deficiency
* Currently smoking tobacco
* Addison's disease
* Allergy to radiographic contrast material
* Symptomatic cholecystolithiasis
* Acute or chronic pancreatitis
* Symptomatic peptic ulcer disease
* Severe unremitting diarrhea, vomiting, or other gastrointestinal disorders that could interfere with the ability to absorb oral medications
* Treatment with antidiabetic medication other than insulin within 4 weeks of enrollment
* Use of any study medication within 4 weeks of enrollment
* Received live attenuated vaccine(s) within 2 months of enrollment
* Any medical condition that, in the opinion of the investigator, might interfere with safe participation

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jose Oberholzer, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Qi M, Kinzer K, Danielson KK, Martellotto J, Barbaro B, Wang Y, Bui JT, Gaba RC, Knuttinen G, Garcia-Roca R, Tzvetanov I, Heitman A, Davis M, McGarrigle JJ, Benedetti E, Oberholzer J. Five-year follow-up of patients with type 1 diabetes transplanted with allogeneic islets: the UIC experience. Acta Diabetol. 2014 Oct;51(5):833-43. doi: 10.1007/s00592-014-0627-6. Epub 2014 Jul 18. PMID 25034311
- [Background] Williams J, Jacus N, Kavalackal K, Danielson KK, Monson RS, Wang Y, Oberholzer J. Over ten-year insulin independence following single allogeneic islet transplant without T-cell depleting antibody induction. Islets. 2018;10(4):168-174. doi: 10.1080/19382014.2018.1451281. Epub 2018 Jul 19. PMID 30024826
- See also: Interest Form — https://uic.ca1.qualtrics.com/jfe/form/SV_1Slg9ZTTfn5zuhE